CLINICAL TRIAL: NCT04936854
Title: Prospective Comparison of Sirolimus Against Corticosteroids in Treatment of Patients With Active Thyroid Eye Disease
Brief Title: Sirolimus vs Corticosteroids in Treatment of Thyroid Eye Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 234527
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Thyroid-Associated Ophthalmopathy
Keywords: Thyroid eye disease; Graves' Orbitopathy; Immunosuppressive Agents; Exophthalmos; Sirolimus
MeSH Terms: conditions — Graves Ophthalmopathy; Exophthalmos | interventions — Sirolimus; Tablets; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant
Masking Description: The treatment will be allocated by the investigator trough the procedure with sealed envelopes, thereafter the investigator will enroll patients and assign patients to treatment. The treatment options will be conceal to prevent participants knowing until final trial analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sirolimus (Active Comparator): Patients with active thyroid eye disease will receive 2 mg Sirolimus (two 1 mg tablets) on the first day, followed by 0,5 mg Sirolimus (half 1 mg tablet) per day for 12 weeks.
  Interventions: Drug: Sirolimus 1 mg Oral Tablet
- Corticosteroids (Active Comparator): Patients with active thyroid eye disease will receive 500 mg Methylprednisolone intravenously once a week for 6 weeks, followed by 250 mg once a week for 6 weeks.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Sirolimus 1 mg Oral Tablet — 2 mg Sirolimus (two 1 mg tablets) on the first day, followed by 0,5 mg Sirolimus (half 1 mg tablet) per day for 12 weeks.
  Other Names: Rapamycin; Rapamune
  Arms: Sirolimus
Drug: Methylprednisolone — 500 mg Methylprednisolone intravenously once a week for 6 weeks, followed by 250 mg once a week for 6 weeks. Total period of treatment 12 weeks.
  Other Names: Solu-Medrol
  Arms: Corticosteroids

SUMMARY:
The purpose of this study is to determine whether Sirolimus is more effective and burdened with less side effects than conventional treatment with corticosteroids in patients with active thyroid eye disease.

DETAILED DESCRIPTION:
Grave's disease is one of the most common autoimmune diseases. Thyroid eye disease is affecting nearly 50% of patients with Grave's disease. European guidelines recommend treating patients with serious TED in the acute face with intravenous steroids for 12 weeks. This treatment is burdened with metabolic complications, like raised blood pressure, high blood glucose, worsening of diabetes, osteoporosis, and weight gain. In addition, peptic ulcer and psychological disturbances are frequently seen. Long-term treatment with high doses of steroids could also suppress the corticotropic axis for a variable time period, giving temporary iatrogenic adrenal insufficiency. It is paramount to develop a treatment with equal or better effect and fewer complications for this group of patients. Recently, Teprotumumab, which act by inhibiting Insulin-Like Growth Factor-1 (IGF-1), has been introduced in treatment of TED. This represents a new area in the anti-inflammatory treatment of the disease. The anti-inflammatory effect of Sirolimus has not been examined in patients with TED, but there are two promising case-reports describing excellent response. Sirolimus have multiple immunosuppressive actions that may be favourable in the inflammatory response in TED. These are: inhibiting T-cell activation, anti-fibroblast effect and blocking the IGF-1 pathway. In contrast to other immunosuppressive drugs, Sirolimus is associated few side effects at low doses.

The investigators are planning a comparative study of conventional treatment (corticosteroids) compared with Sirolimus, regarding clinical outcomes and adverse effects. The investigators plan to include a total of 60 patients (30 in each group) with moderate to severe TED over a period of approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* The participant want treatment for active thyroid eye disease and is willing to be included in the study
* Clinical diagnosis of Graves' disease associated with active TED with a Clinical Activity Score (CAS) ≥ 4 (on the 7-item scale)
* Moderate-to-severe active TED (not sight-threatening but has an appreciable impact on daily life), usually associated with one or more of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, exophthalmos ≥ 3 mm above normal for race and gender, and/or inconstant or constant diplopia
* Onset of active TED symptoms (as determined by participant records) within 9 months prior to inculsion
* Participants must be euthyroid with the Graves disease under control or have mild hypo- or hyperthyroidism (defined as free thyroxine and free triiodothyronine levels < 50% above or below the normal limits).
* Does not require immediate surgical ophthalmological intervention and is not planning corrective surgery/irradiation during the course of the study
* Diabetic participants must have well-controlled stable disease (defined as HbA1C < 9.0% with no new diabetic medication [oral or insulin] or more than a 10% change in the dose of a currently prescribed diabetic medication within 60 days prior to Screening)
* Women of childbearing potential (including those with an onset of menopause <2 years prior to Screening, non-therapy-induced amenorrhea for <12 months prior to Screening, or not surgically sterile [absence of ovaries and/or uterus]) must have a negative serum pregnancy test at Screening and negative urine pregnancy tests at all protocol-specified timepoints (i.e., prior to each dose and through Week 48 of the Follow-Up Period); participants who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the trial, one of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started at least one full cycle prior to Baseline and continue for 180 days after the last dose of study drug. Highly effective contraceptive methods (with a failure rate less than 1% per year) when used consistently and correctly, includes implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence or vasectomized partner
* Male participants must be surgically sterile or, if sexually active with a female partner of childbearing potential, must agree to use barrier contraceptive method from Screening through 180 days after the last dose of study drug
* Active Influenza and Pneumococcal vaccines

Exclusion Criteria:

* The participant dont want treatment for active thyroid eye disease or dont want to participate in the study
* Decreased vision due to optic neuropathy as defined by a significant decrease in best corrected visual acuity, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months
* Corneal decompensation unresponsive to medical management
* Previous orbital irradiation or surgery for TED Any steroid use (intravenous [IV] or oral) with a cumulative dose equivalent to ≥ 1 g of methylprednisolone for the treatment of TED. Previous steroid use (IV or oral) with a cumulative dose of <1 g methylprednisolone or equivalent for the treatment of TED and previous use of steroid eye drops is allowed if the corticosteroid was discontinued at least 4 weeks prior to inclusion
* Corticosteroid use for conditions other than TED within 4 weeks prior to inclusion (topical steroids for dermatological conditions and inhaled steroids are allowed)
* Selenium and biotin must be discontinued 3 weeks prior to Screening and must not be restarted during the clinical trial; however, taking a multivitamin that includes selenium and/or biotin is allowed
* Use of any other non-steroid immunosuppressive including agent, new biologic drugs within 3 months prior to Screening
* Use of an investigational agent for any condition within 60 days prior to inclusion or anticipated use during the course of the trial
* Identified pre-existing ophthalmic disease that, in the judgment of the Investigator, would preclude study participation or complicate interpretation of study results
* Bleeding diathesis that in the judgment of the Investigator would preclude inclusion in the clinical trial
* Malignant condition in the past 12 months (except successfully treated basal/squamous cell carcinoma of the skin)
* Pregnant or lactating women
* Current drug or alcohol abuse, or history of either within the previous 2 years, in the opinion of the Investigator or as reported by the participant
* Biopsy-proven or clinically suspected inflammatory bowel disease
* Known hypersensitivity to any of the components Sirolimus.
* Any other condition that, in the opinion of the Investigator, would preclude inclusion in the study
* Previous enrollment in this study
* Human immunodeficiency virus (HIV), tuberculosis, hepatitis C or hepatitis B infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who were CAS categorical responders at week 12 | Week 12
  CAS categorical responders were defined as participants with a reduction of ≥ 2 CAS points.
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to active (inflammatory phase) thyroid eye disease/ Graves' Ophthalmopathy or Orbitopathy (TED/GO); 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active (inflammatory phase) TED/GO (ignore "equivocal" redness); 6. Chemosis; 7. Inflammation of caruncle or plica. Each item is scored (1=present; 0=absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms).

SECONDARY OUTCOMES:
Percentage of participants who were proptosis responders at week 12 | Week 12
  Proptosis responders were defined as percentage of participants with ≥ 2 mm reduction from baseline in proptosis in one eye at week 12.
Percentage of participants who were eyelid retraction responders at week 12 | Week 12
  Eyelid retraction responders were defined as percentage of participants with ≥ 3 mm reduction from baseline in vertical lid aperture in one eye at week 12
Percentage of participants who were diplopia responders at week 12 | Baseline, up to Week 12
  Diplopia responders were defined as percentage of participants with ≥ 1 class improvement of eye motility from baseline assessed by Gorman score.
  Gorman score: 1 = no diplopia, 2 =intermittent diplopia, 3 = inconstant (gaze-evoked) diplopia, 4 = constant diplopia in primary or reading position.

CONTACTS AND LOCATIONS:
Overall Officials: Hans O Ueland, MD Phd, Principal Investigator — Haukeland University Hospital
Locations (1):
- Department of Ophthalmology Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roos JCP, Murthy R. Sirolimus (rapamycin) for the targeted treatment of the fibrotic sequelae of Graves' orbitopathy. Eye (Lond). 2019 Apr;33(4):679-682. doi: 10.1038/s41433-019-0340-3. Epub 2019 Feb 12. PMID 30755726
- [Background] Chang S, Perry JD, Kosmorsky GS, Braun WE. Rapamycin for treatment of refractory dysthyroid compressive optic neuropathy. Ophthalmic Plast Reconstr Surg. 2007 May-Jun;23(3):225-6. doi: 10.1097/IOP.0b013e3180500d57. PMID 17519662
- [Background] Roos JCP, Eglitis V, Murthy R. Inhibition of Fibrotic Contraction by Sirolimus (Rapamycin) in an Ex Vivo Model of Thyroid Eye Disease. Ophthalmic Plast Reconstr Surg. 2021 Jul-Aug 01;37(4):366-371. doi: 10.1097/IOP.0000000000001876. PMID 33237667